CLINICAL TRIAL: NCT03144258
Title: Evaluation of the Systemic Microcirculation in the Course of Cardiopulmonary Bypass Used in the Surgery for Repair of Congenital Heart Defects in Infants and Children
Brief Title: Evaluation of the Microcirculation During the Corrective Surgery of Congenital Heart Defects in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: CAAE 19201413.6.0000.5272
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart defects; systemic microcirculation; laser Doppler perfusion imaging; cardiac corrective surgery
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
General objective of the research project: To evaluate the alterations of systemic microvascular reactivity during cardiopulmonary bypass (CPB), in children submitted to cardiac surgery for repair of congenital heart defects.

DETAILED DESCRIPTION:
• Specific objectives:

* To test the usefulness of skin laser Doppler flowmetry monitoring (LDPM) in the non-invasive evaluation of endothelium-dependent microvascular reactivity during CPB in children.
* To investigate whether skin LDPM could be proposed as a clinical monitoring of tissue perfusion during CPB in pediatric cardiac surgery.
* To investigate the effects of different anesthetic agents on microvascular reactivity during CPB.
* To investigate the effects of cardiovascular and vasoactive drugs used during CPB on microvascular reactivity.
* To evaluate the correlation of microcirculatory alterations observed during CPB with classical markers of tissue perfusion and oxygenation, including plasma lactate levels.
* To evaluate the correlation of microcirculatory alterations observed during CPB with markers of systemic inflammation, including pro- and anti-inflammatory cytokines.
* To evaluate the correlation of microcirculatory alterations observed during CPB with the plasma bioavailability of nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* infants and children with congenital heart defects scheduled to corrective cardiac surgery

Exclusion Criteria:

* age inferior to 3 months and superior to 6 years

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants and children with congenital heart defects scheduled to corrective cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Microcirculatory alterations during cardiopulmonary bypass | december 2019
  Evaluation of the alterations of microcirculatory parameters and tissue perfusion during cardiopulmonary bypass in children submitted to cardiac corrective surgery for congenital heart defects

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tibirica, MD, PhD, Principal Investigator — National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Ministry of Health, Brazil, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No